CLINICAL TRIAL: NCT03924466
Title: Quantification of 68-GaNOTA-Anti-HER2 VHH1 Uptake in Metastasis of Breast Carcinoma Patients and Assessment of Repeatability (VUBAR) - Pilot Study
Brief Title: Repeatability of 68-GaNOTA-Anti-HER2 VHH1 PET/CT in Breast Carcinoma Patients
Acronym: VUBAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Kom Op Tegen Kanker (Other); Agentschap voor Innovatie door Wetenschap en Technologie, Project Toegepast Biomedisch onderzoek met een primair Maatschappelijke finaliteit. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UZBRU_VHH1_3; 2016-002164-13 (EudraCT Number)
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Breast Carcinoma; Locally Advanced Breast Cancer; Cancer of Pancreas; Solid Tumor With Intermediate or High HER2 Expression; Salivary Gland Cancer; Gastric Cancer; Endometrial Cancer; Uterine Cancer; Non Small Cell Lung Cancer; Biliary Tract Cancer; Cholangiocarcinoma; Colorectal Cancer; Urothelial Carcinoma; Prostate Cancer
Keywords: HER2
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Salivary Gland Neoplasms; Stomach Neoplasms; Endometrial Neoplasms; Uterine Neoplasms; Carcinoma, Non-Small-Cell Lung; Biliary Tract Neoplasms; Cholangiocarcinoma; Colorectal Neoplasms; Carcinoma, Transitional Cell; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial consists of 3 different patient cohorts that are each investigated using a new diagnostic imaging radiopharmaceutical
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients (Experimental): Cohort 1: locally advanced or metastatic breast cancer patients
  Cohort 2: Patients with locally advanced, unresectable, or metastatic cancer disease of breast with low, intermediate or high HER2-expression, salivary gland; gastric body or gastro-esophageal junction; endometrium; uterus; lung; biliary tract; gallbladder; pacreas; colorectum; urothelium; prostate; other solid with intermediate or high HER2-expression
  Cohort 3: Patients with local or locally advanced HER2-+ breast carcinoma, who are planned for neo-adjuvant treatment prior to surgery, and who are suspected for axillary lymph node invasion.
  Interventions: Drug: 68GaNOTA-Anti-HER2 VHH1

INTERVENTIONS:
Drug: 68GaNOTA-Anti-HER2 VHH1 — All subjects will receive at least one single intravenous injection of the IMP followed by a total body PET/CT prior to receiving standard-of-care therapy.
  A second injection of the IMP can be administered before or during standard-of-care treatment, depending on cohort.
  Other Names: HER2-PET/CT

SUMMARY:
Study objective:

Cohort 1: To quantify the uptake of 68GaNOTA-Anti-HER2 VHH1 in local or distant metastases from breast carcinoma patients and to assess repeatability of the image-based HER2 quantification. The uptake will be correlated to results obtained via biopsy of the same lesion, if available.

Cohort 2: To report on uptake of 68GaNOTA-Anti-HER2 VHH1 in different cancer types that might overexpress HER2

Cohort 3: To explore the feasibility and added value of 68GaNOTA-Anti-HER2 VHH1 in the neoadjuvant setting of HER2-expressing breast carcinoma

Time schedule: After inclusion, patients will be injected intravenously with 37 - 185 MBq 68GaNOTA-Anti-HER2 VHH1 with a total mass of up to 200 μg NOTA-Anti-HER2 VHH1. Serum and plasma samples will be collected at injection. At 90 min after injection, a total body PET/CT scan will be performed.

Patients in cohort 1 will undergo a second PET/CT procedure, identical to the first procedure, within 8 days, with a minimal interval of 18h and maximal interval of 8 days. Patients in cohort 2 can undergo an optional 18F-FDG-PET/CT within 21 days prior to or after 68GaNOTA-Anti-HER2 VHH1. In cohort 1 and 2, based on PET/CT images, up to 2 lesions will be selected for optional image-guided biopsy. Biopsy will be performed max. 28 days after the last PET/CT. Plasma and serum samples will be obtained between 60 and 365 days after first injection for patients in cohort 1 and between 42 and 365 days after first injection for patients in cohort 2.

Patients in cohort 3 will undergo 68GaNOTA-Anti-HER2 VHH1 PET/CT prior to the start of neoadjuvant treatment and again after the last cycle of neoadjuvant treatment but prior to surgery. Plasma and serum samples will be obtained before each injection and between 42 and 365 days after the last injection.

ELIGIBILITY:
COHORT SPECIFIC INCLUSION CRITERIA:

COHORT 1:

Patients will only be included in the study if they meet all of the following criteria:

* Patient who has given informed consent
* Patient with age 18 years or older
* Patient with locally or distantly advanced breast carcinoma, with at least 1 lesion of at least 12 mm maximal diameter. For lymph node metastases, the largest diameter should be at least 15 mm and the short axis at least 12 mm.

COHORT 2:

Patients will only be included in the study if they meet all of the following criteria:

* Patient who has given informed consent
* Patient with age 18 years or older
* Patients with locally advanced, unresectable, or metastatic cancer disease , with at least 1 lesion of at least 10 mm maximal diameter (For lymph node metastases, short axis at least 10 mm) of any of the following types:

  * breast carcinoma with low, intermediate or high HER2-expression, based on IHC 1+ or IHC 2+ or IHC 3+, as determined by local assessment on any of the available cancer tissues
  * salivary gland cancer
  * adenocarcinoma of the gastric body or gastro-esophageal junction
  * endometrial cancer
  * cancer of cervix uteri
  * Non-small cell lung cancer
  * biliary tract cancer including intra- or extrahepatic cholangiocarcinoma and tumors arising in the ampulla of Vater or gallbladder.
  * pancreatic cancer
  * colorectal cancer
  * urothelial carcinoma, including transitional cell or predominantly transitional cell carcinoma of the renal pelvis, ureter, urinary bladder or urethra.
  * prostate cancer
  * Other solid malignant tumors with intermediate or high HER2-expression, based on IHC 2+ or IHC 3+, as determined by local assessment on any of the available cancer tissues
* Patients who have progressed following at least one prior systemic treatment for metastatic or advanced disease, or who have no satisfactory alternative treatment option, according to the treating physician (based on all available data such as medical imaging, lab results, clinical examination, …), and who are considered for a next line of systemic treatment. Patients who already participated in the trial and who are diagnosed with progressive or recurrent disease can be re-included if all inclusion criteria and none of the exclusion criteria apply.

COHORT 3:

Patients will only be included in the study if they meet all of the following criteria:

* Patient who has given informed consent
* Patient with age 18 years or older
* Patient with local or locally advanced HER2-positive (either IHC 3+ and/or ISH positive) breast carcinoma, who is planned for neo-adjuvant treatment prior to surgery, and who is suspected for axillary lymph node invasion, based on clinical assessment, ultrasound, CT or MRI, or who has a confirmed lymph node invasion
* Patients who either had 18F-FDG- PET/CT in the last 4 weeks before inclusion, or for whom 18F-FDG- PET/CT is planned before start of neoadjuvant treatment.

GENERAL EXCLUSION CRITERIA:

Patients will not be included in the study if one or more of the following criteria applies:

* Patient is pregnant
* Patient is breast feeding
* Patient with recent (< 1 week) gastrointestinal disorders with diarrhea as major symptom
* Patient with any serious active infection
* Patient who has any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the test radiopharmaceutical
* Patient who cannot communicate reliably with the investigator
* Patient who is unlikely to cooperate with the requirements of the study
* Patient who is unwilling and/or unable to give informed consent
* Patient at increased risk of death from a pre-existing concurrent illness

COHORT SPECIFIC EXCLUSION CRITERIA

COHORT 1 & 3:

* Patient who participated already in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Repeatability of lesional PET/CT characteristics | 90 min post injection
  The lesional tracer uptake in local and distant metastases of at least 12 mm (for lymph nodes short axis) will be measured on both PET/CT's (expressed as standard uptake value (SUV) and repeatability will be calculated.
Tracer update of 68GaNOTA-Anti-HER2 VHH1 in different cancer types | 90 min post injection
  The lesional tracer uptake in different cancer types of at least 10 mm maximal diameter (for lymph nodes short axis) will be measured on PET/CT (expressed as standard uptake value (SUV).
Feasibility and added value of 68GaNOTA-Anti-HER2 in neoadjuvant setting of breast carcinoma | time of surgery following neo-adjuvant treatment (typically within 14 days following the second intervention)

SECONDARY OUTCOMES:
Within-patient tumor heterogeneity for HER2 expression using PET/CT imaging | 90 min post injection
  Within-patient tumor heterogeneity for HER2 expression, observed on 68GaNOTA-Anti-HER2 VHH1 PET/CT or biopsy analyses
Immunogenicity | prior to and between 60 and 365 days after the first injection
  Immunogenicity assessed on plasma samples obtained prior to injection of the IMP and obtained between 60 and 365 days after the (first) injection
Histopathological results of biopsied lesions and correlation with PET/CT results | max 28 days after the second PET/CT
  semi-quantitative score of HER2 expression using immunohistochemistry performed on biopsied/resected tissues if available
Influence image-guide biopsy on patient management | Within 3 months following the last intervention
  To determine in which relative number of patients, the patient management was altered after 68GaNOTA-Anti-HER2 VHH1 PET/CT and the subsequent optional biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Marleen KEYAERTS, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Uz Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No